CLINICAL TRIAL: NCT00280735
Title: Phase II Trial Exploring the Feasibility of Adjuvant Carboplatin/Docetaxel in Curatively Resected Stage I-IIIA Non-Small Cell Lung Cancer
Brief Title: Ph II Adjuvant Carboplatin/Docetaxel in Curatively Resected Stage I-IIIA NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0320
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Trial (Other): adjuvant carboplatin plus docetaxel carboplatin area under curve (AUC) = 6 IV on day 1 every 3 weeks for 4 cycles docetaxel 75 mg/m² IV on day 1 every 3 weeks for 4 cycles
  Interventions: Drug: carboplatin; Drug: docetaxel

INTERVENTIONS:
Drug: carboplatin — Carboplatin will be given intravenously,once,every 3 weeks. The carboplatin area under curve (AUC) dose will be calculated using the Calvert Equation 19 as follows: Carboplatin dose (mg) = 6x (GFR + 25)
  Other Names: paraplatin
Drug: docetaxel — 75 mg/m² intravenously, once, every 3 weeks
  Other Names: Taxotere

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving carboplatin together with docetaxel after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving carboplatin together with docetaxel works in treating patients with stage I, stage II, or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the feasibility of adjuvant carboplatin and docetaxel in patients with resected stage I, II, or IIIA non-small cell lung cancer.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the survival patterns of patients treated with this regimen.
* Assess the patterns of recurrence in patients treated with this regimen.

OUTLINE: Patients receive carboplatin IV on day 1 and docetaxel IV on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed non-small cell lung cancer

  * Stage I-IIIA disease
* Must have undergone a complete resection
* Must begin adjuvant chemotherapy within 8 weeks of surgical resection

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 100,000/mm^3
* Serum creatinine normal OR creatinine clearance ≥ 40 mL/min
* Bilirubin normal
* Alkaline phosphatase (AP), Aspartate aminotransferase (AST), and Alanine transaminase (ALT) must meet 1 of the following criteria:

  * AP normal AND AST and ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST and ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST and ALT normal
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study therapy

Exclusion criteria:

* Patients with a history of severe hypersensitivity to docetaxel or polysorbate 80 are excluded.
* Women who are currently or planning to breast feed.
* Those with peripheral neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

* 2-8 weeks since prior surgery and recovered

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-05 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Socinski, MD, Principal Investigator — Florida Hospital Cancer Institute
Locations (1):
- University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stinchcombe TE, Harper HD, Hensing TA, Moore DT, Crane JM, Atkins JN, Willard EM, Detterbeck FC, Socinski MA. The feasibility of adjuvant carboplatin and docetaxel in patients with curatively resected non-small cell lung cancer. J Thorac Oncol. 2008 Feb;3(2):145-51. doi: 10.1097/JTO.0b013e318160c5f1. PMID 18303435
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 75 participants screened for eligibility, 72 went on to treatment and 3 participants withdrew consent prior to treatment.
Period: Overall Study
Arm/Group | Single Arm Trial
Started | 75
Received Treatment | 72
Received Adequate Exposure (Defined as receiving 4 cycles of therapy within 12 weeks of initiating the first dose.) | 57
Completed | 57
Not Completed | 18
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 8
Not completed — Intercurrent Illness | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 72
Age, Continuous [Median (Full Range); unit: years] | 65 [47 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 68
  Unknown or Not Reported | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 60
  Ethnicity: African American | 7
  Ethnicity: Latino | 2
  Ethnicity: Asian | 1
  Ethnicity: Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 72
Eastern Cooperative Oncology Group (ECOG) Performance status [Count of Participants; unit: Participants] — A scale from 0-5 to describe a patient's level of functioning in terms of selfcare ability and activity level.
  0, Fully active
  1, Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature 2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours 3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours 4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair 5. Dead
  Participants
    0 | 28
    1 | 43
    2 | 1
Stage [Count of Participants; unit: Participants] — Anatomic stage for NSCLC is the American Joint Committee on Cancer (AJCC) tumor node metastatic (TNM) system, which is based on: Size of primary tumor (T) and whether it has grown into nearby areas. Spread to regional lymph nodes (N). Spread (metastasis; M) to other organs of the body. Once the T, N, and M categories have been determined, this information is combined into a prognostic group. Higher numbers mean the cancer is more advanced.
  Participants
    Stage I | 29
    Stage II | 26
    Stage IIIA | 16
    Stage IIIB | 1
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 32
  Squamous cell carcinoma | 30
  Non-small cell-not otherwise specified | 7
  Large cell carcinoma | 3
Type of surgery [Count of Participants; unit: Participants] — Type of pre-screening surgical resection undergone by subjects
  Participants
    Wedge resection | 2
    Lobectomy | 52
    Bi-lobectomy | 7
    Pneumonectomy | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed Four Cycles of the Carboplatin/Docetaxel Regimen
Description: Feasibility was based on the percentage of patients completing four cycles of the carboplatin/docetaxel regimen to a high fraction of patients with curatively resected stage IIIIA non-small cell lung cancer within 12 weeks.
Time Frame: 12 weeks from initiating adjuvant therapy
Population: Patients assigned to treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 72
Participants | 57

2. Secondary Outcome: Patterns of Recurrence in Patients Treated With This Regimen
Description: Patterns were assessed with a staging chest computerized tomography (CT), bone or positron emission tomography (PET) scan and brain magnetic resonance imaging (MRI)/CT scan at recurrence.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm Trial: Patients who relapsed
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 19
Participants
  intrathoracic relapse | 4
  intrathoracic and distant relapse | 5
  distant relapse only without brain | 2
  distant relapse within the brain | 8

3. Secondary Outcome: Toxicity in Patients Treated With This Regimen
Description: Safety determinations are based on the rate of drug-related adverse events (AEs) reported based upon the toxicity as measured by the NCI Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0).
Time Frame: Day 1 of treatment to 30 days after treatment discontinuation
Population: Patients receiving treatment
Measure: Number; unit: percentage of participants
Groups:
- Grade 3 %; Grade 4 %; Grade 3/4 %: Percentage of patients receiving treatment who developed this toxicity
Arm/Group | Grade 3 % | Grade 4 % | Grade 3/4 %
Number analyzed (Participants) | 72 | 72 | 72
percentage of participants
  Neutropenia | 24 | 42 | 65
  Thrombocytopenia | 1 | 0 | 1
  Febrile Neutorpenia | 3 | 8 | 11
  Nausea | 1 | 0 | 1
  Vomiting | 1 | 0 | 1
  Diarrhea | 3 | 0 | 3
  Infusional reactions | 4 | 0 | 4
  Dehydration | 1 | 0 | 1
  Fatigue/asthenia | 5.5 | 0 | 5.5
  Syncope | 5.5 | 0 | 5.5
  Arrythmia | 0 | 1 | 1
  Proteinuria | 0 | 1 | 1
  Infection | 0 | 3 | 3
  Dyspnea | 0 | 1 | 1

4. Secondary Outcome: Progression Free Survival
Description: Relapse-free survival rate at 18 months. Patients were determined to have progression either by radiographic and/or pathological assessment by local physician per local standard of care monitoring for disease recurrence.
Time Frame: The time between the start of treatment to disease progression or death or the date of last contact, measured up to 18 months
Population: Participants receiving treatment
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 72
percentage of participants | 86

5. Secondary Outcome: Overall Survival
Description: Overall survival rate at 18 months.
Time Frame: as for outcome 4
Population: Participants receiving treatment
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 72
percentage of participants | 86

ADVERSE EVENTS:
Time Frame: 30 days following cessation of treatment
Arm/Group | Single Arm Trial
Serious Adverse Events (participants affected / at risk) | 19/72
Other Adverse Events (participants affected / at risk) | 63/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Trial (N=72)
Cardiac ischemia/infarction (Cardiac disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia - Supraventricular arrhythmia not otherwise specified (NOS) (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (9) — Fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infections, Other (Specify, _Neutropenic sepsis) (Infections and infestations) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 2 (3)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 6 (8) — Neutropenia/febrile neutropenia
Leukocytes (total WBC) (Investigations) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Trial (N=72)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 6
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 4
Leukocytes (total WBC) (Investigations) | 4
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 42
Platelets (Investigations) | 1
Supraventricular and nodal arrhythmia - Supraventricular arrhythmia NOS (Cardiac disorders) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 3
Constitutional Symptoms - Other (Specify- Weakness) (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 15
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1
Insomnia (Psychiatric disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 3
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 18
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 9
Heartburn/dyspepsia (Gastrointestinal disorders) | 5
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 13
Taste alteration (dysgeusia) (Nervous system disorders) | 4
Ulcer, GI - Stomach (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Edema: limb (General disorders) | 3
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Mood alteration - Anxiety (Psychiatric disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 3
Syncope (fainting) (Nervous system disorders) | 1
Dry eye syndrome (Eye disorders) | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 2
Pain - bone (Musculoskeletal and connective tissue disorders) | 3
Pain -Chest (General disorders) | 3
Pain - Joint (Musculoskeletal and connective tissue disorders) | 3
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 4
Pain - Other (Specify, _Thoracotomy site) (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other (Specify, _paranasal sinus reaction; runny nose/chills) (Respiratory, thoracic and mediastinal disorders) | 2
Renal/Genitourinary - Other (Specify, __UTI) (Renal and urinary disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days